CLINICAL TRIAL: NCT04704193
Title: Development and Implementation of Electronic Decision Aids for Genetic Testing in Inherited Cancer Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel C Chung, Daniel C Chung, MD; Director, High-Risk GI Cancer Clinic, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P003422; U01CA243695-01 (NIH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Genetic Testing
Keywords: Decision Aid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic Decision Aid (Experimental): Participants in this arm will complete an electronic decision aid for genetic testing.
  Interventions: Other: Survey of Decision Aid

INTERVENTIONS:
Other: Survey of Decision Aid — The decision aid will be evaluated by a survey administered to those who have used the tool.

SUMMARY:
An electronic decision aid will be used to assist individuals in choosing a multi-gene panel with their medical oncologist instead of a genetic counselor. A decision aid may facilitate quality decisions around the selection of a specific multi-gene panel without a genetic counselor. Upon completion of the decision aid, participants will be asked to indicate their decision about whether to pursue genetic testing and which specific multi-gene panel to pursue. A survey will then be administered to assess participants' opinions on the decision aid.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* Diagnosed with malignant ovarian tumor or malignant pancreatic adenocarcinoma

Exclusion Criteria:

* Children (<18 years of age)
* Unable to complete surveys
* Previous germline genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electronic Decision Aid
Started | 93
Completed | 92
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Of the 93 participants, only 92 participants completed the study. Only the information from the 92 participants is included in the baseline characteristics analysis because one participant withdrew from the study.
Arm/Group | Electronic Decision Aid
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 80
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction With How Educational Information is Presented in the Decision Aid
Description: Measured with 6 items on a questionnaire that asks participants to rate the way certain information is presented on the decision aid. Each item is rated on a scale of 1 to 4, with 1 being poor and 4 being excellent.
Time Frame: This outcome will be measured immediately following completion of the decision aid. The average completion time of the decision aid is 14 minutes.
Population: A total of 88 participants agreed to complete this survey. For questions 1b, 1d, and 1e there are only 87 complete answer choices. For question 1f, there are only 86 complete answer choices.
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Decision Aid
Number analyzed (Participants) | 88
Participants
  Genetic testing is a blood test that looks for mutations in genes that can increase cancer risk: Rating: Poor | 1
  Genetic testing is a blood test that looks for mutations in genes that can increase cancer risk: Rating: Fair | 3
  Genetic testing is a blood test that looks for mutations in genes that can increase cancer risk: Rating: Good | 29
  Genetic testing is a blood test that looks for mutations in genes that can increase cancer risk: Rating: Excellent | 55
  Genetic test results may help guide my treatment options: number analyzed (Participants) | 87
  Genetic test results may help guide my treatment options: Rating: Poor | 2
  Genetic test results may help guide my treatment options: Rating: Fair | 4
  Genetic test results may help guide my treatment options: Rating: Good | 30
  Genetic test results may help guide my treatment options: Rating: Excellent | 51
  Genetic test results may help me understand the future risks of other cancers: Rating: Poor | 1
  Genetic test results may help me understand the future risks of other cancers: Rating: Fair | 4
  Genetic test results may help me understand the future risks of other cancers: Rating: Good | 26
  Genetic test results may help me understand the future risks of other cancers: Rating: Excellent | 57
  Genetic test results may increase stress to me and my family members: number analyzed (Participants) | 87
  Genetic test results may increase stress to me and my family members: Rating: Poor | 5
  Genetic test results may increase stress to me and my family members: Rating: Fair | 8
  Genetic test results may increase stress to me and my family members: Rating: Good | 33
  Genetic test results may increase stress to me and my family members: Rating: Excellent | 41
  There are 3 gene panel options that include either a small, medium, or large number of genes: number analyzed (Participants) | 87
  There are 3 gene panel options that include either a small, medium, or large number of genes: Rating: Poor | 2
  There are 3 gene panel options that include either a small, medium, or large number of genes: Rating: Fair | 4
  There are 3 gene panel options that include either a small, medium, or large number of genes: Rating: Good | 31
  There are 3 gene panel options that include either a small, medium, or large number of genes: Rating: Excellent | 50
  Gene test results may come back as positive, negative, or uncertain: number analyzed (Participants) | 86
  Gene test results may come back as positive, negative, or uncertain: Rating: Poor | 1
  Gene test results may come back as positive, negative, or uncertain: Rating: Fair | 6
  Gene test results may come back as positive, negative, or uncertain: Rating: Good | 33
  Gene test results may come back as positive, negative, or uncertain: Rating: Excellent | 46
Statistical Analysis 1: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1a. Genetic testing is a blood test that looks for mutations in genes that can increase cancer risk; Test type: Other — This arm includes descriptive statistics only; count with proportion = .955, 95% CI 2-sided [.888 to .987]
Statistical Analysis 2: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1b. Genetic test results may help guide my treatment options; Test type: Other — This arm includes descriptive statistics only; count with proportion = .931, 95% CI 2-sided [.856 to .974]
Statistical Analysis 3: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1c. Genetic test results may help me understand the future risks of other cancers; Test type: Other — This arm includes descriptive statistics only; count with proportion = .943, 95% CI 2-sided [.872 to .981]
Statistical Analysis 4: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1d. Genetic test results may increase stress to me and my family members; Test type: Other — This arm includes descriptive statistics only; count with proportion = .851, 95% CI 2-sided [.758 to .918]
Statistical Analysis 5: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1e. There are 3 gene panel options that include either a small, medium, or large number of genes; Test type: Other — This arm includes descriptive statistics only; count with proportion = .931, 95% CI 2-sided [.856 to .974]
Statistical Analysis 6: Comparison: Electronic Decision Aid; Descriptive statistics only/proportion reported good or excellent Q1f. Gene test results may come back as positive, negative or uncertain; Test type: Other — This arm includes descriptive statistics only; count with proportion = .919, 95% CI 2-sided [.839 to .967]

2. Secondary Outcome: Total Time Spent on Decision Aid
Description: The total amount of minutes spent on the decision aid
Time Frame: From the start of the decision aid to the completion of the decision aid
Population: There were 85 participants who completed the Electronic Decision Aid tool.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electronic Decision Aid
Number analyzed (Participants) | 85
minutes | 13.7 (5.6)
Statistical Analysis 1: Comparison: Electronic Decision Aid; Test type: Other — Summary statistics only; Mean = 13.7, Standard Deviation 5.6

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Electronic Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT04704193/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04704193/SAP_001.pdf